CLINICAL TRIAL: NCT05357833
Title: Novel Imaging Markers of Innate Immune Activation in Secondary Progressive Multiple Sclerosis
Brief Title: Novel Imaging Markers in SPMS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, M. Mateo Paz Soldan, Assistant Professor, Department of Neurology, Division of Neuroimmunology, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 00147230
Record Dates: First submitted 2022-04-25; First posted 2022-05-03 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Secondary Progressive Multiple Sclerosis; Multiple Sclerosis, Secondary Progressive; Multiple Sclerosis
Keywords: Perilesional microglia; Ferumoxytol; USPIO; Utrasmall superparamagnetic iron oxide nanoparticles; Infiltrating macrophages; Activated microglia; USPIO enhancement
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — Ferrosoferric Oxide; gadoteridol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SPMS Cohort (Experimental): Subjects will undergo MR imaging of the brain and cervical spine for pre- and post-administration of gadoteridol (0.2 mL/kg), then pre- and post-administration of ferumoxytol (4 mg/kg). Scans will be obtained over the course of two separate imaging visits.
  Interventions: Drug: Ferumoxytol infusion; Drug: Gadoteridol; Diagnostic Test: MRI Brain and Cervical Spine

INTERVENTIONS:
Drug: Ferumoxytol infusion — Subjects will receive a single, weighted dose of intravenous ferumoxytol (4 mg/kg) diluted in 50 mL of saline.
  Other Names: Feraheme
Drug: Gadoteridol — Subjects will receive a single, weighted dose of intravenous gadoteridol (0.2 mL/kg).
  Other Names: ProHance, gadolinium-based MRI contrast agent
Diagnostic Test: MRI Brain and Cervical Spine — 3T MR imaging of the brain and cervical spine pre- and post-administration of gadolinium, then pre- and 96 hours (±24 hours) post-administration of ferumoxytol

SUMMARY:
This pilot study takes the innovative approach of using ultrasmall superparamagnetic iron oxide (USPIO) nanoparticle enhanced MRI to measure activity of the innate immune system within MS lesions. Activity of innate immunity has been hypothesized as one of the critical pathologic processes underpinning neurologic worsening in progressive MS. As such, in the short term this project proposes to investigate USPIO uptake in SPMS lesions as a promising in vivo imaging biomarker for chronic-active lesions, as distinguished from chronic-inactive lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 35 to 65 years
2. Clinically diagnosed with secondary progressive multiple sclerosis (SPMS) (2017 McDonald Criteria)
3. Worsening 25 foot walk time (worsening SPMS cohort) over the preceding 2 years.
4. Ambulatory with ability to walk at least 20 meters without rest, with or without aid
5. Ability and willingness to attend study visits and complete the study

Exclusion Criteria:

1. Clinically diagnosed with relapsing remitting multiple sclerosis (RRMS), primary progressive multiple sclerosis (PPMS), clinical isolated syndrome (CIS), or radiologically isolated syndrome (RIS)
2. Clinical MS relapse and/or new MRI lesion(s) within the preceding 2 years
3. Positive pregnancy test
4. Gadolinium contrast allergy
5. Acute or chronic kidney disease with eGFR <30 ml/min/1.73m2
6. Pacemaker or other MRI contraindications per American College of Radiology guidelines
7. Intravenous iron sensitivity
8. Serum ferritin and transferrin saturation above age-adjusted upper limit of normal (if serum ferritin is above normal, but transferrin saturation is normal, the subject is NOT excluded)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Signal change on T1-weighted and 3D UTE MRI brain (and upper cervical cord) before and 96 hours (±24 hours) after ferumoxytol administration | 96 hours ±24 hours

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability) | 96 hours ±24 hours
  Assess the safety and tolerability of ferumoxytol in Secondary Progressive MS cohort based on Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: M. Mateo Paz Soldan, MD, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Imaging and Neurosciences Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No